CLINICAL TRIAL: NCT01718600
Title: Long-term Neurocognitive Sequelae of Subclinical Microembolization During Carotid Interventions
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University of Wisconsin, Madison (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: R01NS070308 (NIH)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery stenting; neuropsychological testing; microembolization; MRI
MeSH Terms: conditions — Carotid Stenosis | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Neuroimaging Correlates: Carotid revascularization can significantly reduce the risk of stroke in patients with severe carotid stenosis; however, it has been associated with cognitive decline in 25% of the older adults who undergo the procedure. Neuroimaging techniques that characterize white matter integrity and regional hypoperfusion have the potential to provide sensitive brain structure indicators that may be associated with memory decline following revascularization procedures. In this proposal, we hope to determine the risk factors and cognitive effect of microembolization following carotid revascularization procedures.
  Interventions: Behavioral: Neuropsychological testing

INTERVENTIONS:
Behavioral: Neuropsychological testing

SUMMARY:
Microembolization is commonly associated with carotid artery stenting (CAS), but our understanding of subclinical microembolization is superficial. Through collaborative effects of multidisciplinary team-experts, novel approaches, and longitudinal evaluations, we hope to better understand the clinical significance and long-term cognitive effects of microemboli. This proposal may change our current clinical practice by providing a better outcome measure for carotid interventions and improving outcomes of CAS procedures through risk factor stratification. Our central hypothesis is that development of subclinical microemboli is associated with decline in cognitive function following CAS and that the risk of development of microemboli themselves is associated with patient- and procedure-related factors. We hope that this prospective study will help to clarify these important issues in the era of rapidly evolving percutaneous interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female >40 yrs of age.
* Patient has occlusive extracranial carotid stenosis (≥70%)
* Patient is scheduled to undergo an endovascular intervention of a lesion in the extracranial carotid artery
* Patient agrees to voluntarily participate and signs an informed consent.
* Patient agrees to be available for follow-up and is able to participate in all study testing procedures.
* Patient has sufficient visual and auditory acuity for cognitive testing.

Exclusion Criteria:

* Patient is unable to safely and comfortably undergo magnetic resonance imaging procedures (e.g., claustrophobia, implanted medical devices that are MRI incompatible such as pacemaker, defibrillator, neural stimulator etc)
* Patient has an untreated or unsuccessfully controlled psychiatric disease (schizophrenia, bipolar disorder).
* Patient has prominent suicidal or homicidal ideation.
* Patient has acute illness or unstable chronic illness (e.g. uncontrolled hypertension, hepatic encephalopathy, portal hypertension, ascites, and esophageal varices, pancreatitis).
* Patient with a history of neurological (e.g., multiple sclerosis, seizure disorder, Parkinson's disease) or systemic illness affecting central nervous system function.
* Patient has prior closed head injury with ≥24 hours of amnesia.
* Patient is unable to understand or sign the informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing carotid intervention
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Incidence of microemboli in correlation with changes in neurocognitive assessment performance | 1 year following CAS procedure

SECONDARY OUTCOMES:
Risk factor stratification for incidence of microemboli | 1 year following CAS procedure

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Palo Alto Veterans Affairs, Palo Alto, California
  - Washington University School of Medicine, St Louis, Missouri
  - University of Wisconsin, Madison, Madison, Wisconsin

REFERENCES:
- [Background] Zhou W, Hitchner E, Gillis K, Sun L, Floyd R, Lane B, Rosen A. Prospective neurocognitive evaluation of patients undergoing carotid interventions. J Vasc Surg. 2012 Dec;56(6):1571-8. doi: 10.1016/j.jvs.2012.05.092. Epub 2012 Aug 11. PMID 22889720